CLINICAL TRIAL: NCT03341988
Title: Evaluation of the Clinical Effects of Ombitasvir/Paritaprevir/Ritonavir Regimen in the Treatment of Chronic HCV Patients in CKD Versus ESRD Patients in Assiut University Hospital
Brief Title: Evaluation of Treatment of Chronic HCV Patients in Chronic Kidney Disease Versus End Stage Renal Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed A Mekky, Clinical professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCV in renal impairment
Record Dates: First submitted 2017-10-02; First posted 2017-11-14 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ombitasvir (25 mg ), Paritaprevir (150 mg ) once daily (Other): Ombitasvir (25 mg once daily), Paritaprevir (150 mg once daily), Ritonavir (100 mg once daily)Ribavirin (RBV): weight-based and divided bid (1000 mg/day if < 75kg or 1200 mg/day if ≥ 75kg) given to 50 chronic HCV infected patients with renal impairment for 12 week
  Interventions: Drug: Ombitasvir-Paritaprevir-Ritonavir Tab 12.5-75-50 milligram

INTERVENTIONS:
Drug: Ombitasvir-Paritaprevir-Ritonavir Tab 12.5-75-50 milligram — To asses curability of( Ombitasvir ,Paritaprevir,Ritonavir) in ch HCV infected patients in those with CKD vs ESRD 2- Also assess duration of sustained viral response,treatment, relapse or failure of therapy in CKD vs ESRD

SUMMARY:
1. To asses curability of( Ombitasvir ,Paritaprevir,Ritonavir) in chronic HCV infected patients in those with CKD versus ESRD in Assiut Hospital University .
2. Also assess duration of sustained viral response,treatment, relapse or failure of therapy in CKD versus ESRD in Assiut Hospital.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a leading cause of liver disease worldwide, as 130-170 million individuals are chronically infected and 350,000 patients die every year from HCV infection. The HCV prevalence varies widely among countries being highest in several African and Eastern Mediterranean countries. So public health authorities should recognise the importance of HCV and make resources available for the implementation of effective primary prevention, screening and management policies .

The hepatitis C virus (HCV) genotype is an important predictor of disease progression and treatment response. Genotype 1b has a worldwide distribution and is often found to be the most common genotype. HCV-genotype 4 causes approximately 20% of the 180 million cases of chronic hepatitis C in the world, is predominant in the Middle East and Northern Africa, and has recently spread to Southern Europe. Genotype 4 accounts for more than 90% of the reported cases from Egypt, a country with a massive HCV-related disease burden.

The prevalence of anti-hepatitis C virus Ab (anti-HCV) positivity among dialysis patients varies across countries, ranging from 3 to 75%; unfortunately, Egypt is considered one of the countries with the highest prevalence despite the existence of guidelines for a comprehensive infection control program.

In Egypt In the 15-59-year age groups, the prevalence of HCV antibody was found to be 10.0% and that of HCV RNA to be 7.0%. Approximately, 3.7 million persons have chronic HCV infection in the age group 15-59 in 2015.

In the treatment of chronic HCV in renal impairment For patients with mild to moderate renal impairment (CrCl 30 mL/min-80 mL/min), no dosage adjustment is required when using fixed-dose combination of paritaprevir (150 mg)/ritonavir (100 mg)/ombitasvir (25 mg) .

Abbvie's 2D regimen (paritaprevir (150 mg)/ritonavir (100 mg)/ombitasvir(25mg)) was recently approved with specific indication for genotype 4 treatment naïve and experienced patients without cirrhosis achieved an sustained viral response rate of 100% following 12 weeks of 2D regimen with RBV, 2D can be used without RBV but may have slightly lower SVR (91% vs 100%). Currently, there is no FDA indication for 2D regimen use in patients with cirrhosis.

. Ombitasvir (25 mg once daily), Paritaprevir (150 mg once daily), Ritonavir (100 mg once daily)Ribavirin (RBV): weight-based and divided bid (1000 mg/day if < 75kg or 1200 mg/day if ≥ 75kg) .

ELIGIBILITY:
Inclusion Criteria:

1. The patients aged from18- 60 years.
2. Chronic HCV infection with Plasma HCV RNA greater than 15,000 IU/mL
3. Treatment naïve.
4. compensated liver cirrhosis.
5. Absence of coinfection with HBV or HIV.

Exclusion Criteria:

1. Patients with hepatitis B virus or HIV.
2. prior antiviral therapy.
3. Haemoglobin level less than 10mg/dl.
4. Decompensated liver disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the sustained viral response of Ombitasvir/Paritaprevir/Ritonavir regimen in the treatment of Chronic HCV patients in CKD versus ESRD patients in Assiut University Hospital | 6 months
  pathologic complete remission for HCV after tretment

CONTACTS AND LOCATIONS:
Overall Officials: Hala Elsherif, Professor, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Hezode C, Asselah T, Reddy KR, Hassanein T, Berenguer M, Fleischer-Stepniewska K, Marcellin P, Hall C, Schnell G, Pilot-Matias T, Mobashery N, Redman R, Vilchez RA, Pol S. Ombitasvir plus paritaprevir plus ritonavir with or without ribavirin in treatment-naive and treatment-experienced patients with genotype 4 chronic hepatitis C virus infection (PEARL-I): a randomised, open-label trial. Lancet. 2015 Jun 20;385(9986):2502-9. doi: 10.1016/S0140-6736(15)60159-3. Epub 2015 Mar 31. PMID 25837829
- [Background] Zhang J, Nguyen D, Hu KQ. Chronic Hepatitis C Virus Infection: A Review of Current Direct-Acting Antiviral Treatment Strategies. N Am J Med Sci (Boston). 2016 Apr;9(2):47-54. Epub 2016 Apr 27. PMID 27293521
- [Background] Kandeel A, Genedy M, El-Refai S, Funk AL, Fontanet A, Talaat M. The prevalence of hepatitis C virus infection in Egypt 2015: implications for future policy on prevention and treatment. Liver Int. 2017 Jan;37(1):45-53. doi: 10.1111/liv.13186. Epub 2016 Jun 30. PMID 27275625
- [Derived] Mekky MA, Abdel-Malek MO, Osman HA, Abdel-Aziz EM, Hashim AA, Hetta HF, Morsy KH. Efficacy of ombitasvir/paritaprevir/ritonavir/ribavirin in management of HCV genotype 4 and end-stage kidney disease. Clin Res Hepatol Gastroenterol. 2019 Feb;43(1):82-87. doi: 10.1016/j.clinre.2018.08.003. Epub 2018 Aug 27. PMID 30166253